CLINICAL TRIAL: NCT01991093
Title: The Role of Multiple Electrode Aggregometry in Detection of Clopidogrel Resistance in Diabetic Patients With Coronary Artery Disease and Prediction of Clinical Outcomes. A Comparative-method, Non Interventional, Single Center Study.
Brief Title: Multiple Electrode Aggregometry & Clopidogrel Resistance
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013-11-IIS
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Coronary Artery Disease (CAD); Myocardial Infraction
Keywords: light transmittance aggregometry (LTA),multiple electrode aggregometry, clopidogrel-resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Antiplatelet therapy with aspirin-clopidogrel reduces the risk of cardiovascular episodes after percutaneous coronary intervention (PCI) in patients with acute coronary syndromes. However, a significant number of patients experience recurrent events while on such therapy. The individual response to dual antiplatelet therapy is not uniform, and consistent findings across multiple investigations support the association between a lower degree of platelet inhibition, high on-treatment platelet reactivity, and the occurrence of atherothrombotic events [1, 2]. Particularly in diabetic patients, clopidogrel resistance is more prevalent compared with non-diabetics [3,4], which seems to contribute to the increased atherothrombotic risk in these patients compared with those without diabetes mellitus (DM) [5]. A number of platelet function instruments have now become available that are simple to use and can be utilized as point-of-care (POC) instruments in order to monitor antiplatelet therapy and potentially assess the risk of a recurrent event [6].

DETAILED DESCRIPTION:
The aim of this study is to evaluate the ability of a new POC device, the multiple electrode aggregometry (Multiplate, Dynabyte, Munich, Germany) to detect clopidogrel resistance and predict the clinical outcome in patients with type 2 diabetes mellitus (T2DM) and coronary artery disease (CAD) in comparison with the light transmittance aggregometry (LTA), which is considered the gold standard of platelet function testing [7]. 280 patients with T2DM between 20 and 75 years of age treated with oral and/or parenteral hypoglycaemic therapy for at least 1 month and angiographically established coronary artery disease on the grounds of a previous ST elevation, non-ST elevation acute coronary syndrome or unstable angina treated with clopidogrel 75 mg/day in combination with daily per os aspirin therapy for at least 7 days after documentation of CAD, will be recruited. Patients' enrollment will take place in the Second University Department of Cardiology of the "Attiko" University Hospital in Athens, Greece. Baseline assessment will include recording of demographic data, medical history, cardiovascular risk factors, hematological parameters, number of diseased vessels, number of stented vessels, previous myocardial infarction (MI), previous revascularization, ejection fraction and concomitant medications. Patients with renal (creatinine levels > 2.5 mg/dl) or hepatic (bilirubin level > 2 mg/dL) insufficiency, malignant disease, use of drugs known to affect platelet function, history of bleeding diathesis, platelet count < 100x109/L and a hematocrit < 28% will be excluded. The protocol will be approved by the institutional review board of "Attiko" University Hospital and all patients will give written informed consent before undergoing any study procedure or receiving any study treatment.

Platelet function measurements will be performed on study enrollment. Patients will be identified either as poor or good responders to clopidogrel. The primary end-point will be defined as a composite of death from cardiovascular causes, nonfatal myocardial infarction, stent thrombosis, ischemic stroke, urgent rehospitalization for acute coronary syndrome and/or revascularisation during 1-year follow-up period. Episodes of major bleeding according to PLATO criteria will be recorded during follow-up [8].

The ability of the two methods to detect clopidogrel resistance will be evaluated and the potential correlation between response to antiplatelet treatment and clinical outcome will be assessed. In parallel, patients with similar characteristics, but treated with prasugrel or ticagrelor, will be used as control group of the same sample size.

Platelet Function Analysis Platelet function analysis will be performed in the Laboratory of Haematology and Blood Bank Unit of "Attiko" University Hospital. Blood samples will be collected from an antecubital vein 2 to 4 h after antiplatelet therapy intake. The first 2 to 4 ml of blood will be discarded to avoid spontaneous platelet activation and platelet function tests will be performed within two hours of sampling.

Light transmittance aggregometry (LTA) The whole blood specimen will be collected in 3.8% trisodium citrate and centrifuged at 200 g for 10 minutes to obtain platelet-rich plasma (PRP). The remaining specimen will be re-centrifuged at 2000 g for 15 minutes to obtain platelet-poor plasma (PPP). The platelet count will be adjusted to between 200,000/μl and 300,000/μl with PPP. Aggregation will be performed using a Biodata-PAP-4 aggregometer (Bio/Data Corporation, PA, USA). The 100% line will be set using PPP and a 0% baseline established with PRP before addition of the agonist. The agonist used will be ADP 2.0×10-5 M (Bio/Data Corporation, PA, USA). Test procedure will be performed as previously described [9]. In brief, 0.45 mL PRP is transferred into a cuvette incubated at 37 °C for 3 minutes. Then 0.05 mL of the agonist is added into the PRP and the aggregation pattern is allowed to generate for 6 minutes. Platelet aggregation was determined as the maximal percent change in light transmittance from baseline using PPP as a reference. Cut-off value of > 59% aggregation following 20 microM ADP stimulation will be defined as that indicating of high on-treatment platelet reactivity [10]. Other tested parameters will be late aggregation and the degree of disaggregation.

Multiple electrode aggregometry (MEA) Platelet aggregation in whole blood will be assessed by MEA using an impedance aggregometer (Multiplate, Dynabyte, Munich, Germany). Samples will be collected into 3.2% citrate tubes and analyzed within the period of half to two hours after blood collection according to manufacturer's instructions. Platelet aggregation will be induced by ADP in final concentration 6.5 μM. Each disposable test cell contains two pairs of electrodes, thus enabling two simultaneous measurements. Aggregation will reported as area under the curve (AUC), an integrated measure of aggregation velocity and maximal aggregation. Cut-off value for HRPR by MEA (> 468 arbitrary aggregation units/min in response to ADP by Multiplate analyzer) was defined according to the recently published consensus statement on the definition of high on-treatment platelet reactivity to adenosine diphosphate [11].

Statistical Methods

1. Primary endpoint:

   In this prospective cohort study, the primary end point will be defined as a composite of death from cardiovascular causes, nonfatal myocardial infarction, stent thrombosis, ischemic stroke, urgent rehospitalisation for acute coronary syndrome and/or revascularisation during the 1-year follow-up period. Episodes of major bleeding according to PLATO criteria will be recorded during follow-up.
2. Descriptive statistics:

   They will be presented as means ± SD, medians and interquartile ranges (IQR), or percentages when appropriate.
3. Comparison of baseline data (demographic data, medical history, cardiovascular risk factors, hematological parameters, number of diseased vessels, previous myocardial infarction, previous revascularisation, ejection fraction and concomitant medications) between responders and non-responders to clopidogrel:

   First, we will use the Shapiro-Wilk test to check for the normality of data distributions. Continuous variables will be compared by means of the two-sample Student's t test (when the distribution is found normal) or by means of the non-parametric two-sample Wilcoxon rank-sum (Mann-Whitney) test (when the distribution is found non-normal). Categorical variables will be compared using the Pearson's chi-squared test.
4. Agreement of the two methods in detecting resistance to clopidogrel:

   Agreement between "Multiplate" and "ADP-induced LTA" will be determined by kappa statistics and the respective p-values. Kappa values of < 0.20 are considered to indicate poor agreement, 0.21 to 0.40 indicate fair agreement, 0.41 to 0.60 indicate moderate agreement, 0.61 to 0.80 indicate good agreement, and >0.81 indicate very good agreement.
5. Correlation of laboratory resistance with clinical outcome:

   Logistic regression analysis will be used in order to evaluate whether the methods of detecting resistance to clopidogrel ("Multiplate" and "ADP-induced LTA") are associated with the clinical outcome (end-point). To evaluate whether these associations are independent, certain covariates that are well-known risk factors (ie., cardiovascular risk factors, number of diseased vessels, previous myocardial infarction, previous revascularisation, etc) will be included in the multivariable logistic regression models. The crude and the adjusted odds ratios (ORs) and the corresponding 95% confidence intervals (CIs) will be presented.
6. Level of significance:

   For hypothesis testing, a probability level of < 0.05 will be considered as statistically significant. All statistical tests will be two-sided.
7. Statistical software:

   Stata software will be used for all statistical analyses (Stata Corp., College Station, TX, USA).
8. Sample size calculation:

For the study sample size calculation, we hypothesize that clopidogrel resistance CR(+) is more prevalent among T2DM patients compared with non-DM patients [12, 13]; at the same time, the DM group of patients with clopidogrel resistance suffer an increased likelihood of adverse cardiovascular events [14]. It has been shown that 13% of the general population of T2DM patients suffer a major adverse cardiovascular event (MACE) [including death secondary to cardiovascular cause, ST-segment elevation myocardial infarction (STEMI), non-ST-segment elevation myocardial infarction (NSTEMI) and unstable angina (UA) and stroke]; this number increases to 38% among T2DM patients with clopidogrel resistance who remain on clopidogrel treatment [15]. The sample size needed to detect this difference in adverse event rates - between CR(+) and CR(-) diabetic patients - with a two-sided a risk of 5% and a b risk of 20% (power of 80%) will have to be 101 patients [40 in CR(+) group and 61 in CR(-) group]. If we assume an attrition rate of 10%, the sample size should be further increased to 111 patients [44 in CR(+) group and 67 in CR(-) group]. Finally, taking under consideration that clopidogrel resistance among T2DM patients can be estimated to reach approximately 40% [16-18], the initial sample of all diabetic patients should be 2.5 times larger, or 278 patients (111 clopidogrel-resistant and 167 clopidogrel-sensitive). The statistical software G*Power 3.1.3 (Kiel, Germany) was used for sample size calculation.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus (T2DM)
* coronary artery disease (CAD)patients
* males and females
* patients who will be on clopidogrel treatment
* patients treated with prasugler or ticagrelor after an ACS will also undergo platelet reactivity tests, will be followed-up to record the primary endpoint for one year and will serve as control group to patients treated with clopidogrel
* patients who will sign the study informed consent form
* patients who will comply with all study procedures

Exclusion Criteria:

* patients who will not sign the study informed consent form
* patients who will not comply with all study procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes mellitus (T2DM) and coronary artery disease (CAD)patients who will be detected for clopidogrel resistance
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Multiple electrode aggregometry in detection of clopidogrel resistance | 7 days
  Percentage of type 2 diabetes mellitus (T2DM) and coronary artery disease (CAD)patients who are detected as clopidogrel resistance and predict the clinical outcome in comparison with the light transmittance aggregometry (LTA), which is considered the gold standard of platelet function testing

CONTACTS AND LOCATIONS:
Overall Officials: Argirios Tsantes, MD, Ass Professor, Study Chair — Head of Laboratory of Haematology & Blood Bank Unit, "Attiko" University General Hospital
Locations (3):
- Greece (3):
  - 2nd Cardiology Department,, Athens, Haidari, Athens
  - Attikon University Hospital, Athens, Haidari
  - Laboratory of Haematology & Blood Bank Unit, "Attiko" University General Hospital, Athens

REFERENCES:
- [Background] Geisler T, Langer H, Wydymus M, Gohring K, Zurn C, Bigalke B, Stellos K, May AE, Gawaz M. Low response to clopidogrel is associated with cardiovascular outcome after coronary stent implantation. Eur Heart J. 2006 Oct;27(20):2420-5. doi: 10.1093/eurheartj/ehl275. Epub 2006 Sep 27. PMID 17005534
- [Background] Sibbing D, Braun S, Morath T, Mehilli J, Vogt W, Schomig A, Kastrati A, von Beckerath N. Platelet reactivity after clopidogrel treatment assessed with point-of-care analysis and early drug-eluting stent thrombosis. J Am Coll Cardiol. 2009 Mar 10;53(10):849-56. doi: 10.1016/j.jacc.2008.11.030. PMID 19264241
- [Background] Angiolillo DJ, Fernandez-Ortiz A, Bernardo E, Ramirez C, Sabate M, Jimenez-Quevedo P, Hernandez R, Moreno R, Escaned J, Alfonso F, Banuelos C, Costa MA, Bass TA, Macaya C. Platelet function profiles in patients with type 2 diabetes and coronary artery disease on combined aspirin and clopidogrel treatment. Diabetes. 2005 Aug;54(8):2430-5. doi: 10.2337/diabetes.54.8.2430. PMID 16046311
- [Background] Geisler T, Anders N, Paterok M, Langer H, Stellos K, Lindemann S, Herdeg C, May AE, Gawaz M. Platelet response to clopidogrel is attenuated in diabetic patients undergoing coronary stent implantation. Diabetes Care. 2007 Feb;30(2):372-4. doi: 10.2337/dc06-1625. No abstract available. PMID 17259513
- [Background] Angiolillo DJ. Antiplatelet therapy in diabetes: efficacy and limitations of current treatment strategies and future directions. Diabetes Care. 2009 Apr;32(4):531-40. doi: 10.2337/dc08-2064. No abstract available. PMID 19336638
- [Background] Price MJ. Bedside evaluation of thienopyridine antiplatelet therapy. Circulation. 2009 May 19;119(19):2625-32. doi: 10.1161/CIRCULATIONAHA.107.696732. No abstract available. PMID 19451364
- [Background] Harrison P, Frelinger AL 3rd, Furman MI, Michelson AD. Measuring antiplatelet drug effects in the laboratory. Thromb Res. 2007;120(3):323-36. doi: 10.1016/j.thromres.2006.11.012. Epub 2007 Jan 17. PMID 17239428
- [Background] James S, Akerblom A, Cannon CP, Emanuelsson H, Husted S, Katus H, Skene A, Steg PG, Storey RF, Harrington R, Becker R, Wallentin L. Comparison of ticagrelor, the first reversible oral P2Y(12) receptor antagonist, with clopidogrel in patients with acute coronary syndromes: Rationale, design, and baseline characteristics of the PLATelet inhibition and patient Outcomes (PLATO) trial. Am Heart J. 2009 Apr;157(4):599-605. doi: 10.1016/j.ahj.2009.01.003. PMID 19332184
- [Background] Tsantes AE, Dimoula A, Bonovas S, Mantzios G, Tsirigotis P, Zoi K, Kalamara E, Kardoulaki A, Sitaras N, Travlou A, Dervenoulas J, Vaiopoulos G. The role of the Platelet Function Analyzer (PFA)-100 and platelet aggregometry in the differentiation of essential thrombocythemia from reactive thrombocytosis. Thromb Res. 2010 Feb;125(2):142-6. doi: 10.1016/j.thromres.2009.06.030. Epub 2009 Aug 7. PMID 19664802
- [Background] Gurbel PA, Antonino MJ, Bliden KP, Dichiara J, Suarez TA, Singla A, Tantry US. Platelet reactivity to adenosine diphosphate and long-term ischemic event occurrence following percutaneous coronary intervention: a potential antiplatelet therapeutic target. Platelets. 2008 Dec;19(8):595-604. doi: 10.1080/09537100802351065. PMID 19012177
- [Background] Bonello L, Tantry US, Marcucci R, Blindt R, Angiolillo DJ, Becker R, Bhatt DL, Cattaneo M, Collet JP, Cuisset T, Gachet C, Montalescot G, Jennings LK, Kereiakes D, Sibbing D, Trenk D, Van Werkum JW, Paganelli F, Price MJ, Waksman R, Gurbel PA; Working Group on High On-Treatment Platelet Reactivity. Consensus and future directions on the definition of high on-treatment platelet reactivity to adenosine diphosphate. J Am Coll Cardiol. 2010 Sep 14;56(12):919-33. doi: 10.1016/j.jacc.2010.04.047. PMID 20828644
- [Background] Angiolillo DJ, Bernardo E, Ramirez C, Costa MA, Sabate M, Jimenez-Quevedo P, Hernandez R, Moreno R, Escaned J, Alfonso F, Banuelos C, Bass TA, Macaya C, Fernandez-Ortiz A. Insulin therapy is associated with platelet dysfunction in patients with type 2 diabetes mellitus on dual oral antiplatelet treatment. J Am Coll Cardiol. 2006 Jul 18;48(2):298-304. doi: 10.1016/j.jacc.2006.03.038. Epub 2006 Jun 22. PMID 16843179
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Angiolillo DJ, Bernardo E, Sabate M, Jimenez-Quevedo P, Costa MA, Palazuelos J, Hernandez-Antolin R, Moreno R, Escaned J, Alfonso F, Banuelos C, Guzman LA, Bass TA, Macaya C, Fernandez-Ortiz A. Impact of platelet reactivity on cardiovascular outcomes in patients with type 2 diabetes mellitus and coronary artery disease. J Am Coll Cardiol. 2007 Oct 16;50(16):1541-7. doi: 10.1016/j.jacc.2007.05.049. Epub 2007 Oct 1. PMID 17936152
- [Background] Angiolillo DJ, Shoemaker SB, Desai B, Yuan H, Charlton RK, Bernardo E, Zenni MM, Guzman LA, Bass TA, Costa MA. Randomized comparison of a high clopidogrel maintenance dose in patients with diabetes mellitus and coronary artery disease: results of the Optimizing Antiplatelet Therapy in Diabetes Mellitus (OPTIMUS) study. Circulation. 2007 Feb 13;115(6):708-16. doi: 10.1161/CIRCULATIONAHA.106.667741. Epub 2007 Jan 29. PMID 17261652
- [Background] Erlinge D, Varenhorst C, Braun OO, James S, Winters KJ, Jakubowski JA, Brandt JT, Sugidachi A, Siegbahn A, Wallentin L. Patients with poor responsiveness to thienopyridine treatment or with diabetes have lower levels of circulating active metabolite, but their platelets respond normally to active metabolite added ex vivo. J Am Coll Cardiol. 2008 Dec 9;52(24):1968-77. doi: 10.1016/j.jacc.2008.07.068. PMID 19055987
- [Background] Angiolillo DJ, Badimon JJ, Saucedo JF, Frelinger AL, Michelson AD, Jakubowski JA, Zhu B, Ojeh CK, Baker BA, Effron MB. A pharmacodynamic comparison of prasugrel vs. high-dose clopidogrel in patients with type 2 diabetes mellitus and coronary artery disease: results of the Optimizing anti-Platelet Therapy In diabetes MellitUS (OPTIMUS)-3 Trial. Eur Heart J. 2011 Apr;32(7):838-46. doi: 10.1093/eurheartj/ehq494. Epub 2011 Jan 20. PMID 21252171